CLINICAL TRIAL: NCT06038721
Title: Unified Protocol: Community Connections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Children's Trust, Miami FL (Other)
Responsible Party: Principal Investigator, Jill May Ehrenreich, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230860
Record Dates: First submitted 2023-09-07; First posted 2023-09-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Issue; Anxiety Disorder; Depressive Disorder; Parenting
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Children (Experimental): The participants in this group will receive the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Children (UP-C) in up to 15 sessions through a group format, attended over up to 24 weeks. Sessions will include parent and child strategies to manage strong emotions.
  Interventions: Behavioral: The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Children
- The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Adolescents (Experimental): The participants in this group will receive the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) in an individual format for up to 24 weeks.
  Interventions: Behavioral: The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Adolescents

INTERVENTIONS:
Behavioral: The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Children — The UP-C is administered in-person to parents and children over the course of up to 15 weekly group sessions, which last approximately 90 minutes each.
  Other Names: UP-C
  Arms: The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Children
Behavioral: The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Adolescents — The UP-A is administered to parents and teens over the course of approximately 15-24 weekly individual sessions, which last approximately 50 minutes each. Sessions can be administered in-person or online, with at least one session occurring in person.
  Other Names: UP-A
  Arms: The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Adolescents

SUMMARY:
The purpose of this study is to administer the Unified Protocols for Transdiagnostic Treatment of Emotional Disorders in Children (UP-C) and Adolescents (UP-A) to youth and participants' parents and to examine the efficacy and outcomes of the treatment using standardized measures, questionnaires, interviews. The UP-C and the UP-A are cognitive-behavioral therapies to treat emotional disorders.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 7-17.
* Youth currently resides in Miami-Dade County.
* Children and their parents must be able to speak and understand English and/or Spanish sufficiently well to complete study procedures (e.g., provide their informed consent/assent, complete assessment measures and/or program materials).
* At least one parent or caregiver with whom the child is living with that can accompany the child and participate in all visits (assessment and treatment).
* Positive endorsement of elevated emotional concerns in one of a limited range of emotional disorder domains (i.e., anxiety, depression, trauma, or obsessive-compulsive symptoms, etc.) during full DIAMOND-Kid semi-structured interview, and/or elevated anxiety or depression symptoms (T-Score > or = 65 for youth 8-17 years old; Raw score > or = 12 for children under 8 years old) on the Revised Child Anxiety and Depression Scale - Short Form (RCADS-SF; Child or Parent Report).
* Youth with other types of comorbid conditions (e.g., tic/Tourette's disorder, eating disorders, or disruptive behavior disorders) will not be excluded, providing a clinical area of concern is regarding one of the emotional disorder domains specified and treatment within this protocol is deemed most appropriate.
* Youth and parent participation in at least one in-person session if the treatment is predominantly delivered virtually.

Exclusion Criteria:

* Prior receipt of at least 8 sessions of the UP-C/A program at the Child and Adolescent Mood and Anxiety Treatment Program (CAMAT).
* Psychiatric hospitalization in the previous 6 months (i.e., due to Baker Act, psychotic symptoms, significant suicidal ideation, danger to self or others, etc.).
* Another significant problem area that takes priority for services (e.g., eating disorder, substance-use disorder, primary externalizing concerns, psychotic symptoms, etc.), as identified by family report or via DIAMOND-Kid interview.
* Inability for family to wait for the next group treatment cohort to start, family declining therapist assignment following intake, and/or family no-showing to 3 or more scheduled sessions at CAMAT (inclusive of intake assessment).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-25 (Estimated)

PRIMARY OUTCOMES:
Change in Revised Children's Anxiety and Depression Scale - Parent Revised Short Version (RCADS-P-S) | Session 1 (approximately week 1), session 8 (approximately week 8), and at the natural termination session (approximately 24 weeks).
  The Change in Revised Children's Anxiety and Depression Scale - Parent Revised Short Version (RCADS-P-25) is 25-item parent-reported scale measuring symptoms of anxiety and depression in youth. Items are rated on a 4-point scale from 1 (Never) to 4 (always) with total composite score ranging from 0 to 75. A score of 70 or higher indicates high severity.
Change in Revised Children's Anxiety and Depression Scale - Child Revised Short Version (RCADS-C-S) | Session 1 (approximately week 1), session 8 (approximately week 8), and at the natural termination session (approximately 24 weeks).
  The Change in Revised Children's Anxiety and Depression Scale - Child Revised Short Version (RCADS-25) is 25-item self-reported scale measuring symptoms of anxiety and depression in youth. Items are rated on a 4-point scale from 1 (Never) to 4 (always) with total composite scores ranging from 0 to 75. A score of 70 or higher indicates high severity.
Change in Strengths and Difficulties Questionnaire - Parent Version (SDQ-P) | Session 1 (approximately week 1), session 8 (approximately week 8), and at the natural termination session (approximately 24 weeks).
  The Strengths and Difficulties Questionnaire (SDQ) is a 25-item parent-reported measure assessing five domains in youth: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and pro-social behaviors. All items are rated on a 3-point scale from 0 (not true) to 2 (Certainly true). A score can be generated for each scale and all except the prosocial subscale are added together to generate a total composite difficulties score (based on 20 items). Higher total scores are indicative of more problems for all subscales, except for the prosocial scale, where higher scores correspond to fewer difficulties in prosocial behavior.
Change in Strengths and Difficulties Questionnaire - Child Version (SDQ-C) | Session 1 (approximately week 1), session 8 (approximately week 8), and at the natural termination session (approximately 24 weeks).
  The Strengths and Difficulties Questionnaire (SDQ) is a 25-item self-reported measure assessing five domains in youth: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and pro-social behaviors. All items are rated on a 3-point scale from 0 (not true) to 2 (Certainly true). A score can be generated for each scale and all except the prosocial subscale are added together to generate a total composite difficulties score (based on 20 items). Higher total composite scores are indicative of more problems for all subscales, except for the prosocial scale, where higher scores correspond to fewer difficulties in prosocial behavior.
Change in Parental Stress Scale (PSS) as measured by Likert Scale | Session 1 (approximately week 1), session 8 (approximately week 8), and at the natural termination session (approximately 24 weeks).
  The Parental Stress Scale (PSS) is an 18-item measure assessing parents' feelings about their parenting role, exploring both positive (e.g., emotional benefits, personal development) and negative (e.g., demands on resources, feelings of stress) aspects on parenthood. All items are rated on 5-point Likert scale from 1 (Strongly disagree) to 5 (Strongly agree). Items are summed with higher scores indicating higher levels of parental stress.

SECONDARY OUTCOMES:
Top Problems Assessment - Parent Report as measured by Likert Scale | up to 24 weeks
  The Top Problems assessment is used to identify parent-reported target problems for treatment and track changes in problem severity over time. Identified top problem statements are rated on 9-point Likert scale from 0 (not at all a problem) to 8 (a huge problem).
Top Problems Assessment - Child Report as measured by Likert Scale | up to 24 weeks
  The Top Problems assessment is used to identify self-reported target problems for treatment and track changes in problem severity over time. Identified top problem statements are rated on 9-point Likert scale from 0 (not at all a problem) to 8 (a huge problem).
Change in Clinical Global Impression, Severity Scale (CGI-S) | At baseline, and up to 24 weeks
  The CGI-S is a single-item clinician-reported measure used to assess the severity of the youth's illness at the time of assessment. The item is rated on a 7-point scale ranging from 1 (very much improved since the initiation of treatment) to 7 (very much worse since the initiation of treatment). Higher scores indicate greater symptom severity.
Clinical Global Impression - Improvement (CGI-I) | At up to 24 weeks
  The CGI-I is a single-item clinician-reported measure used to assess clinical changes in youth symptomology over the course of treatment. The item is rated on a 7-point scale ranging from 1 (very much improved since the initiation of treatment) to 7 (very much worse since the initiation of treatment). Higher scores indicate greater symptom improvement since baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ehrenreich-May, PhD, Principal Investigator — University of Miami
Locations (1):
- Child and Adolescent Mood and Anxiety Treatment Program, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehrenreich-May, J., Kennedy, S. M., Sherman, J. A., Bilek, E. L., Buzzella, B. A., Bennett, S. M., & Barlow, D. H. (2017). Unified protocols for transdiagnostic treatment of emotional disorders in children and adolescents: Therapist guide. Oxford University Press.